CLINICAL TRIAL: NCT06832761
Title: Secondary Prevention of Dementia in Memory Clinics: Implementation and (Cost-)Effectiveness of an Integrated Lifestyle Intervention
Brief Title: Lifestyle Intervention in the Memory Clinics of General and Academic Hospitals Trial
Acronym: LIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); InHolland University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL86513.068.24; 10930012310012 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-12-23; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Lifestyle Intervention; Lifestyle Risk Reduction; Cognitive Decline; Dementia
Keywords: Lifestyle intervention; Risk reduction; Dementia; Memory clinic
MeSH Terms: conditions — Risk Reduction Behavior; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: Group A receives a personalised lifestyle intervention. Group B will receive general information on lifestyle in relation to dementia risk reduction.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle intervention (Group A) (Experimental): Group A receives a personalized lifestyle intervention.
  Interventions: Behavioral: Personalized lifestyle intervention
- Regular healthcare (Group B) (No Intervention): Group B receives regular health care and a folder with general information on lifestyle and dementia risk reduction.

INTERVENTIONS:
Behavioral: Personalized lifestyle intervention — The lifestyle intervention in Group A comprises three parts (1) three individual consultations with a trained lifestyle coach, (2) a voucher program to encourage brain healthy activities, and (3) access to an online self-management tool for dementia risk reduction (www.breinzorg.nl).
  Arms: Lifestyle intervention (Group A)

SUMMARY:
Lifestyle Intervention in the memory clinics of General and academic Hospitals Trial (LIGHT) is a multi-center, randomized, controlled, lifestyle intervention trial among 300 older adults (≥50 years) with subjective cognitive decline (SCD) and mild cognitive impairment (MCI) at risk of dementia. Participants are randomized in a 1:1 ratio to Group A (tailored lifestyle intervention) or Group B (general health advice) for a duration of 12 months. The lifestyle intervention comprises three parts 1) Lifestyle coaching, 2) a voucher program, and 3) online self-management. Group B will receive general health advice.

DETAILED DESCRIPTION:
Rationale: Dementia prevention through lifestyle has much potential but is not implemented in routine care. Patients referred to memory clinics, such as people with mild cognitive impairment (MCI) and subjective cognitive disorder (SCD), are at high risk for dementia and tend to have a worse health and lifestyle profile. While they might greatly benefit from lifestyle changes, there is no offer to help them make those changes.

Objective: The primary objectives are to examine both the (cost-)effectiveness of an innovative 1-year lifestyle intervention on lifestyle change measured by the validated Lifestyle for Brain Health Score (LIBRA) in older adults with SCD or MCI; and to identify possibilities, barriers, and facilitators for sustainable implementation of the lifestyle intervention.

Study design: Multicenter, randomized controlled trial comparing a lifestyle intervention with care as usual and general health advice.

Study population: 300 older adults (≥50 years) with SCD and MCI at risk of dementia.

Intervention: Participants are randomly allocated on a 1:1 ratio to participate either in Group A (tailored lifestyle intervention) or Group B (general health advice) for a duration of 12 months. The lifestyle intervention comprises three parts 1) Lifestyle coaching, 2) a voucher program, and 3) online self-management. Group B will receive general health advice.

Main study parameters/endpoints: The primary outcome will be change in participants' dementia risk profile as measured by the LIBRA score between baseline and 12 months. Secondary outcomes include cognitive functions (episodic memory, executive functions, information processing speed and attention). Other secondary outcomes include measures of body mass index (height and weight), office systolic and diastolic blood pressure, and lab measures including cholesterol levels (total, HDL, LDL, triglycerides), HbA1c levels, creatinine-based eGFR levels. Smoking, alcohol intake and current relevant medical conditions (coronary heart disease, kidney disease, type 2 diabetes, depression, hearing loss, sleep disorders) will be assessed through self-report. Additional questionnaires include health-related quality of life and capabilities, instrumental activities of daily living, health locus of control, self-efficacy, mastery, healthy diet, physical activity, cognitive stimulation, stress, and depressive symptoms, sleep quality, social support and feelings of loneliness, and lastly knowledge on dementia risk and protective factors. For cost-effectiveness, questionnaires on resource utilization, medical consumption, and productivity costs are administered. Additional measures include change in diagnosis (if applicable), demographics (age, sex, educational level, socioeconomic position (household income), paid/voluntary work hours, ethnicity, marital status, living situation), medication use, hearing loss. For process evaluation, questionnaires and interviews are administered on implementation, mechanisms of impact and contact (e.g., appointments with lifestyle coach, use of the breinzorg.nl self-management tool, use of the voucher program, experiences and usefulness, etc.).

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age at pre-screening;
* Having a diagnosis of SCD or MCI;
* Presence of ≥ 2 modifiable risk factors for dementia.

Exclusion Criteria:

* Having a diagnosis of dementia;
* Insufficient understanding of the Dutch language;
* Conditions affecting safe and continuous engagement in the intervention (e.g. under treatment for current malignant diseases, major psychiatric disorders (e.g. major depression, psychosis, bipolar disorder), other conditions preventing co-operation as judged by the local study nurse or consulted physician at the local study site;
* Participation in any other research intervention trial at time of pre-screening and throughout the study period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Lifestyle for BRAin Health (LIBRA) score 2 | 1 year
  1-year change in the Lifestyle for BRAin Health (LIBRA) score 2. This is a weighted score of fifteen lifestyle-related risk factors that are proven to be associated with increased dementia risk. Higher score means a greater risk for dementia. Scored from -6.1 to 25.8 (absolute weight).

SECONDARY OUTCOMES:
15-Word Verbal Learning Test | 1 year
  Measure of immediate and delayed memory. Wordlist is presented five times in a row and asked to be recalled immediately and after 15 minutes.
  Discrete number; score: 0-15 (higher score means a better outcome)
Digit Symbol Substitution Test (DSST) | 1 year
  Measure of attention/processing speed, number of correctly matched symbols to digits within 90 seconds.
  Discrete number; 0-90 (higher score means a better outcome).
Wechsler Adult Intelligent Scale (WAIS) digit span | 1 year
  Measure of working memory. Scored as the maximum number of digits repeated correctly. Discrete number; 0-14 (higher score means a better outcome).
Trail Making Test | 1 year
  Measure of attention and executive function. Task A and B. Time taken to complete the test; minimum 0, no maximum, lower score means a better outcome.
Semantic Fluency Test | 1 year
  Measure of language fluency. Semantic fluency test with category animals at baseline and professions at follow-up. Word count in one minute; minimum 0, no maximum, higher score means a better outcome.
EuroQol-5D-5L | 1 year
  Quality of life, score 0-100, higher scores indicate better quality of life
ICEpop CAPability measure for Older people (ICECAP-O) | 1 year
  Capabilities, score 0-1, higher scores indicate greater capabilities.
Health locus of Control Scale | 1 year
  3 subscales, where each subscale ranges from 6 (minimum score) to 36 (maximum score). Higher scores indicate higher health locus of control.
General Self-Efficacy scale | 1 year
  Total score ranges from 10 (minimum score) to 40 (maximum score), with higher scores representing higher self-efficacy.
Pearlin Mastery Scale | 1 year
  Total score ranges from 7 (minimum score) to 28 (maximum score), where higher scores indicate greater levels of mastery.
Cholesterol | 1 year
  Total, HDL, LDL and triglycerides in plasma (mmol/L).
Hemoglobin A1c | 1 year
  Hemoglobin A1C (HbA1c) measured in plasma (%), indicates plasma glucose as a measure for diabetes status
Estimated glomerular filtration rate (eGFR) | 1 year
  Creatinine-based (as measured in plasma) estimated glomerular filtration rate (eGFR) (healthy level: higher than 60) indicating kidney function.
Body mass Index (BMI) | 1 year
  As calculated from weight (kg) and height (m), weight / height ^2
Blood pressure | 1 year
  Scores range from approximately (for diastolic) 60-120 and (for systolic) 100-180 mmHg, with higher measures indicating higher blood pressure.
Medical history | 1 year
  History of diabetes, coronary heart disease, kidney disease, hypertension, dyslipidemia, depression, hearing loss, poor vision, sleep disorders (asked in interview)
Amsterdam-Instrumental Activities Daily Living (ADL) Questionnaire | 1 year
  Total scores range approximately 20-70, higher scores indicate better ADL functioning.
Mediterranean Diet Adherence Screener (MEDAS) | 1 year
  Total score ranges from 0 (minimum score) to 14 (maximum score), with higher scores indicating higher adherence to Mediterranean diet.
Investigation into Cancer and Nutrition (EPIC) physical activity questionnaire | 1 year
  Physical activity, uses Cambridge Physical Activity Index to categorize into 4 levels based on occupational and leisure-time activities.
Cognitive and Leisure Activities Scale | 1 year
  The score ranges from 0 (minimum score) to 45 (maximum score), with higher scores representing higher cognitive and leisure activities.
Perceived Stress Scale | 1 year
  Total score, scale 0 - 40, higher scores indicate more perceived stress.
Patient Health Questionnaire (PHQ)-9 | 1 year
  Total score ranges from 0 (minimum score) to 27 (maximum score), with higher scores representing a worse outcome (more depressive symptoms).
Groningen Sleep Quality Scale (GSKS) | 1 year
  The score ranges from 0 (minimum score) to 14 (maximum score), with higher scores representing a worse outcome (worse sleep quality)
6-item Lubben social network Scale | 1 year
  The score ranges from 0 (minimum score) to 30 (maximum score), with higher scores meaning a better outcome (higher level of perceived social support)
De Jong Gierveld 6-item Scale | 1 year
  The score ranges from 0 (minimum score) to 6 (maximum score), with higher scores representing a worse outcome (higher loneliness scores).
Knowledge on dementia risk questionnaire | 1 year
  Measure awareness on risk and protective factors, higher score indicates better knowledge (0-25).
Smoking | 1 year
  Duration (current/history) and quantity
Alcohol intake | 1 year
  Measured in duration (current/history) and quantity
Medical Consumption Questionnaire (iMCQ) | 1 year
  Medical consumption, selection of specific questions on care use such as GP visits and dietician. Used to calculate overall costs of medical care to define the cost-effectiveness of the intervention. Lower costs is a better score.
Productivity Costs Questionnaire (iPCQ) | 1 year
  Measures productivity costs, used to calculate cost-effectiveness of the intervention. Higher productivity and lower costs is a better score.
Adherence | 1 year
  Appointments missed, personal goals reached in coaching sessions (number), vouchers used (number), usage log of breinzorg.nl self-management tool (time active, modules completed). Together, they will be used in a model to calculate cost-effectiveness of the intervention based on the adherence.

OTHER OUTCOMES:
Biomarkers | 1 year
  Plasma samples will be stored to later assess biomarkers. For example amyloid, p-tau, NFL, GFAP, BDNF.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Köhler, Professor, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Alzheimer Center Amsterdam, Amsterdam
  - Maastricht University, Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deckers K, Zwan MD, Soons LM, Waterink L, Beers S, van Houdt S, Stiensma B, Kwant JZ, Wimmers SCPM, Heutz RAM, Claassen JAHR, Oosterman JM, de Heus RAA, van de Rest O, Vermeiren Y, Voshaar RCO, Smidt N, Broersen LM, Sikkes SAM, Aarts E; MOCIA consortium; FINGER-NL consortium; Kohler S, van der Flier WM. A multidomain lifestyle intervention to maintain optimal cognitive functioning in Dutch older adults-study design and baseline characteristics of the FINGER-NL randomized controlled trial. Alzheimers Res Ther. 2024 Jun 13;16(1):126. doi: 10.1186/s13195-024-01495-8. PMID 38872204
- [Background] Rosenau C, Kohler S, Soons LM, Anstey KJ, Brayne C, Brodaty H, Engedal K, Farina FR, Ganguli M, Livingston G, Lyketsos CG, Mangialasche F, Middleton LE, Rikkert MGMO, Peters R, Sachdev PS, Scarmeas N, Salbaek G, van Boxtel MPJ, Deckers K. Umbrella review and Delphi study on modifiable factors for dementia risk reduction. Alzheimers Dement. 2024 Mar;20(3):2223-2239. doi: 10.1002/alz.13577. Epub 2023 Dec 30. PMID 38159267
- [Derived] van Gils V, Waterink L, Wimmers SCPM, Jelsma JGM, de Vugt ME, Handels R, Sikkes SAM, van der Flier WM, Deckers K, Zwan MD, Kohler S, Janssen N. The Lifestyle Intervention in memory clinics of General and academic Hospitals Trial (LIGHT): Rationale and study design of a randomized controlled trial to reduce modifiable dementia risk. Alzheimers Res Ther. 2026 Jan 8;18(1):31. doi: 10.1186/s13195-025-01947-9. PMID 41508135
- See also: ZonMw description — https://projecten.zonmw.nl/nl/project/dementierisico-reductie-individueel-leefstijladvies-de-leefstijl-interventie-op-de
- See also: Alzheimer Center Limburg description — https://www.alzheimercentrumlimburg.nl/light